CLINICAL TRIAL: NCT01829867
Title: A Phase I, Open-label Study in Patients With Parkinson's Disease to Further Assess Safety and Tolerability of sNN0031 Administered at the Total Dose of 95 μg by Intracerebroventricular Infusion
Brief Title: A Study With an Increased Dose Step in Patients That Have Previously Received Placebo or sNN0031.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues with development and supply of infusion system for delivery of IMP. Prolonged approval process for the clinical study sNN0031-004.
Sponsor: Newron Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sNN0031-003
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sNN0031 (Experimental)
  Interventions: Drug: sNN0031

INTERVENTIONS:
Drug: sNN0031

SUMMARY:
The purpose of this study is to assess the safety and tolerability of a dose of 95μg sNN0031 after intracerebroventricular administration to patients with Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of idiopathic PD
* Previous participation in study sNN0031-001 with completion of 12 study weeks without development of clinically significant safety concerns defined as being any drug-related or device related SAE that resulted in premature termination of treatment or a medical device incident that could not be resolved during the conduct of study sNN0031-001 and sNN0031-002
* Inclusion in study sNN0031-002 and participation without development of clinically significant safety concerns defined as being device related SAE that resulted in premature termination or a medical device incident that could not be resolved during the conduct of study sNN0031-002
* Intact continuity of the SynchroMed® II pump and ICV-catheter infusion system as judged by X-ray of head and abdominal area
* An ICV catheter tip position that is similar to the catheter tip position at implantation in study sNN0031-001, as verified with an MRI not older than 3 months
* Verification of device function made as a comparison of pump actual residual volume to the anticipated residual volume as indicated by the programmer. Reference point will be the refill volume and programming of the pump made at first visit with saline refill in study sNN0031-002. Values within 25% of expected will be an indication that the pump is functioning properly
* Ophthalmologic examination with no clinically significant findings that imply safety concerns for this study such as retinal haemorrhage, signs for papillary oedema
* Females should either be post-menopausal (at least 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhoea with follicle stimulating hormone levels >40 mIU/mL), be surgically sterilised (bilateral oophorectomy without hysterectomy), or use adequate contraception (oral contraceptives, intrauterine device or double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam) during the duration of the study
* The patient, with or without the help of a caregiver, must be capable of maintaining an accurate and complete symptom diary and to adhere to visit schedules
* The patient has been given written and verbal information about the study, has had the opportunity to ask questions about the study, and understands the time and procedural commitments
* The patient has provided written informed consent to participate in the study before any study-specific procedures are conducted

Exclusion Criteria:

* Participation in another clinical study that entails investigational drug or device treatment after participation in study sNN0031-001 or study sNN0031-002
* The patient has, since participation in study sNN0031-001, had functional neurosurgical treatment for PD (e.g., deep brain stimulation)
* Concurrent dementia with a score of 20 or lower on the MoCA-test
* Concurrent clinically significant depression with a score of 16 or higher on the MADRS rating scale, equivalent to moderate or severe depression.
* Exposure to neuroleptic drugs blocking dopamine receptors within 6 months from the baseline visit of this study
* History of structural brain disease including tumours and hyperplasia
* Ongoing or suspected primary or recurrent malignant disease
* History of increased intracranial pressure
* Uncontrolled hypertension with blood pressure >160 mmHg systolic or >90 mmHg diastolic.
* Completion of an MRI examination of the brain and cervical spinal cord within 3 months prior to study start with finding of tumours or potential sources of pathological bleedings, or abnormality that may or would interfere with the assessments of safety or efficacy, in the judgment of the Investigator
* Presence of cardiac pacemakers, spinal cord stimulators, implantable programmable intraspinal drug pumps, or any other device that may interfere or interact with the programmer
* Clinically significant abnormalities in haematology or clinical chemistry parameters indicative of a medical condition requiring treatment which, in the opinion of the Investigator, is not compatible with participation in the present study
* Ongoing medical condition that according to the Investigator would interfere with the conduct and assessments in the study. Examples are medical disability (e.g., severe degenerative arthritis, compromised nutritional state, peripheral neuropathy) that would interfere with the assessment of safety and efficacy of investigational product or device performance, or would compromise the ability of the patient to undergo study procedures (e.g., MRI), to maintain a patient diary or to give informed consent.
* Serological evidence of HBV, HCV or HIV.
* Tuberculosis (TB) as detected by positive findings in chest X-ray and microscopy of urine.
* Increased susceptibility to infections (e.g. malignancies, neutropenia, immunodeficient states, immunosuppressive therapy).

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events per participant | 12 months

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) parts I, II and III | Change from baseline to 6 months
Quality of Life assessed by the use of the EQ-5D | "Change from baseline to 6 months" and "Change from baseline to 12 months"
Montgomery-Åsberg Depression Rating Scale (MADRS) | "Change from baseline to 3 months" and "Change from baseline to 6 months" and "Change from baseline to 12 months"
Montreal Cognitive Assessment (MoCA) | "Change from baseline to 3 months" and "Change from baseline to 6 months" and "Change from baseline to 12 months"

CONTACTS AND LOCATIONS:
Overall Officials: Gesine Paul-Visse, Principal Investigator — Skånes University Hospital Lund
Locations (2):
- Sweden (2):
  - Skåne University Hospital Lund, Lund
  - Karolinska University Hospital Huddinge, Stockholm